CLINICAL TRIAL: NCT01195116
Title: Usefulness of Dexmedetomidine on Post-operative Pain Management in Patients With Interstitial Cystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Suzanne Karan, Principal investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB 31154
Record Dates: First submitted 2010-08-13; First posted 2010-09-03 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Interstitial Cystitis
Keywords: Post-operative pain management; Pain Management; Painful bladder syndrome; frequency and urgency; Dexmedetomidine; hydrodistension
MeSH Terms: conditions — Cystitis, Interstitial; Agnosia | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine is a FDA-approved medication that is a highly selective, short acting, alpha-2 adrenoreceptor agonist. To date, its safety and efficacy is well studied and established.It produces sedative, anxiolytic, and analgesic effects when used while patients undergo procedures and surgical operations.Interstitial Cystitis, as a chronic visceral pain syndrome, has the potential to have a neuropathic component for which an alpha-2 adrenergic agonist may be more effective than other classes, including opioids or NSAIDs.
  Interventions: Drug: Dexmedetomidine
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — 1 mcg/kg/hour
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Normal Saline — 1mcg/kg/hr
  Other Names: Sodium Chloride
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to assess the effects of dexmedetomidine while patients undergo treatment for Interstitial Cystitis (IC). The investigators goal is to demonstrate in patients with IC undergoing bladder hydrodistension that the use of dexmedetomidine as a supplemental anesthetic agent will result in better postoperative pain management.

DETAILED DESCRIPTION:
Inclusion Criteria: Patients with a clinical diagnosis of IC scheduled for cystoscopy and hydrodistension for both diagnostic and therapeutic indications.

Data collected will include:

I. Postoperative Outcomes i. Pain Reported (Visual Analogue Scale) ii. Post-operative opiate use iii. Time in PACU iv. Time until discharge v. Adverse Events (i.e. nausea/vomiting, nursing intervention) II. Intermediate-term Outcomes (4-6 weeks) i. Interstitial Cystitis Symptom & Problem Index ii. Revised McGill Pain Score

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of IC scheduled for cystoscopy and hydrodistension for both diagnostic and therapeutic indications.
* 2. Gender of Patients: Male & female,Age of Patients: 18 and older

Exclusion Criteria:

* Conduction disturbance (second degree AV block or greater), or previous reaction to medications used in this study. Patients receiving spinal anesthesia will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Karan, MD, Principal Investigator — University of Rochester Department of Affiliation; Robert Mayer, MD, Principal Investigator — University of Rochester Department of Urology; Denham Ward, MD, PhD, Principal Investigator — University of Rochester Department of Anesthesiology
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Normal Saline
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: subjects were recruited if they were scheduled for bladder lavage under general anesthesia for the treatment of interstitial cystitis
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Normal Saline | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.32 (10.98) | 45.25 (15.25) | 47 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score (1-10, 10 is Most Pain) From Baseline, to Average Post op Pain Score in PACU
Description: It is a measurement instrument for subjective characteristics or attitudes towards pain that cannot be directly measured.
Time Frame: Assessed every 15 minutes while in Post Anesthesia Care Unit until discharged home, which was approximately 10 times on the average
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Normal Saline
Number analyzed (Participants) | 21 | 20
units on a scale | -1.46 (3.33) | -.025 (4.88)

ADVERSE EVENTS:
Arm/Group | Dexmedetomidine | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No